CLINICAL TRIAL: NCT06038513
Title: A Prospective, Open Label Clinical Trial to Evaluate the Safety and Efficacy of the COOLSTAT® Transnasal Thermal Regulating Device in Inducing Normothermia for Neurogenic Fever in an Intensive Care Setting
Brief Title: Transnasal Induction of Normothermia for Neurogenic Fever
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: CoolTech LLC (Industry)
Collaborators: Maryland Industrial Partnerships (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COT-002
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Seizures; Metabolic Encephalopathy
Keywords: shivering, fever, normothermia, TTM
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Seizures; Brain Diseases, Metabolic; Fever; Trichotillomania

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transnasal Thermal Regulating Device (Experimental): Consented subjects who develop fever will undergo cooling via transnasal thermal regulating device for a period of 24 hours
  Interventions: Device: Transnasal Thermal Regulating Device

INTERVENTIONS:
Device: Transnasal Thermal Regulating Device — Placement of transnasal thermal regulating device to reduce temperature in febrile patients for a period of 24 hours
  Other Names: CoolStat

SUMMARY:
The objective of this study is to evaluate the efficacy of the COOLSTAT® Transnasal Thermal Regulating Device in reducing temperature in a population of febrile subjects who meet the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to an Intensive Care Unit for a planned stay of at least 24 hours with a diagnosis of ischemic or hemorrhagic stroke, seizure, or metabolic encephalopathy.
2. Ages 18-85 years, inclusive.
3. Patient has fever ≥ 38.3°C and ≤ 38.9°C at the time of treatment initiation.
4. Patient is orally intubated or has tracheostomy tube and is mechanically ventilated.
5. Glasgow Coma Scale score of 3-11, inclusive.
6. Must have informed consent from the patient or the legally authorized representative (LAR) making decisions for the patient.

Exclusion Criteria:

1. Intubation is contraindicated.
2. Weight of ≤ 100lb or ≥ 250lb.
3. Active/ongoing epistaxis.
4. Known or suspected pregnancy.
5. Participation in another ongoing investigational study.
6. Prisoners and/or patients for whom no LAR is available.
7. Patient is in airborne/droplet disease isolation protocol.
8. Patient is or suspected to be immunocompromised.
9. Nasal septal deviations (per standard of care CT scan; any degree).
10. Chronic rhinosinusitis.
11. Traumatic brain injury.
12. Prior skull-base surgery.
13. Penetrating cranial trauma.
14. Recent nasal trauma or anterior base skull fracture.
15. Any condition for which transnasal air flow would be contraindicated.
16. Refractory hypoxemia (partial pressure of oxygen in arterial blood (paO2) below 60 torr or oxyhemoglobin saturation below 90% despite endotracheal intubation, mechanical ventilation, and provision of supplemental oxygen of up to 0.60).
17. Refractory hypercarbia (partial pressure of carbon dioxide in arterial blood (paCO2) above 50 torr despite endotracheal intubation and conventional mechanical ventilation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Time to achieve normothermia (≤37.5°C) | 24 hours
  To evaluate the efficacy of the COOLSTAT® in reducing temperature in a population of febrile subjects who meet the inclusion/exclusion criteria.

SECONDARY OUTCOMES:
Temperature burden above 37.5°C (°C*hours) during the 24-hour cooling period | 24 hours
  To evaluate the efficacy of the COOLSTAT® in maintaining normothermia over a 24-hour cooling period
Incidence of shivering during cooling period | 24 hours
  To assess the frequency of shivering incidents caused by the CoolStat device.
Number of shivering interventions per patient | 24 hours
  To assess the frequency shivering interventions caused by the CoolStat device.
Incidence of adverse events. | 24 hours
  To evaluate the safety of the CoolStat device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No